CLINICAL TRIAL: NCT00783497
Title: Stress, Blood Pressure, & Ethnicity
Brief Title: Evaluating the Relationship Between Stress, Ethnicity, and Blood Pressure
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joel E. Dimsdale, M.D., Emeritus Professor, University of California, San Diego
Other Study IDs: 599; R01HL036005 (NIH); 5R01HL036005-23 (NIH)
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Stress
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Caucasian Americans
- 2: African Americans

SUMMARY:
High blood pressure is a common health problem among people in the United States. This study will examine the ways that stress and ethnicity play a role in the development of high blood pressure.

DETAILED DESCRIPTION:
High blood pressure affects nearly one third of all people in the United States. It can be caused by many factors, including obesity, sodium intake, genetics, and stress. Ethnicity appears to also play a role, because African Americans are more susceptible to developing high blood pressure than other ethnic groups, with more than 40% of African Americans diagnosed with this condition. This study will examine the underlying reasons of why stress and African-American ethnicity contribute to high blood pressure risk and how ethnicity and stress interact with each other to increase this risk. Specifically, study researchers will examine how stress increases blood pressure, how people from different ethnic groups respond to stress differently, and how sleep plays a role in regulating blood pressure levels.

This study will enroll African Americans and Caucasians who have high blood pressure, as well as African Americans and Caucasians who have normal blood pressure. Potential participants will go through a screening process that involves a medical history review, questionnaires, and blood pressure monitoring. Eligible participants will then be admitted to the research clinic for a 2-night stay. Participants' nutrition history and body measurements will be obtained, and a catheter will be inserted into the arm so that blood can be easily collected during the clinic stay. During the night, participants' breathing habits and movements will be monitored while they sleep. During the day, blood pressure and heart activity will be monitored frequently, including when participants are asked to perform mildly stressful tasks, such as giving a short speech. Various medications that affect heart rate and blood pressure will be given at different times during the study, and researchers will monitor participants' reactions to each medication. Lastly, participants will also complete psychological questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as African American or Caucasian
* Weighs 85% to 150% of ideal weight (approximate BMI of 17.5 to 30)
* In good physical health

Exclusion Criteria:

* Blood pressure greater than 180/110 mm Hg at any point in the past
* Currently works less than half-time
* Currently is employed doing shift work
* Currently takes prescription medication, other than anti-hypertensive medication
* Currently smokes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample in the San Diego, California metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2005-10; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel E. Dimsdale, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States